CLINICAL TRIAL: NCT00988780
Title: CCR5 Antagonism to Decrease the Incidence of the Immune Reconstitution Inflammatory Syndrome in HIV-Infected Patients
Brief Title: Maraviroc (CCR5) Antagonism to Decrease the Incidence of the Immune Reconstitution Inflammatory Syndrome in HIV-Infected Patients
Acronym: CADIRIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: University of Witwatersrand, South Africa (Other); Case Western Reserve University (Other); The Wistar Institute (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Juan G. Sierra Madero, Infectious Diseases Specialist, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: The CADIRIS Study
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Immune Reconstitution Inflammatory Syndrome; HIV; HIV Infections
Keywords: Immune reconstitution inflammatory syndrome; CCR5 antagonist; Maraviroc; HIV; treatment naive
MeSH Terms: conditions — Immune Reconstitution Inflammatory Syndrome; HIV Infections | interventions — Maraviroc; efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maraviroc (Experimental): Maraviroc 600mg po BID
  Background antiretroviral regimen (Efavirenz 600mg QD + Tenofovir 300 mg /Emtricitabine 200 mg QD) plus Maraviroc 600 mg BID
  Interventions: Drug: maraviroc
- Placebo (Placebo Comparator): Placebo po BID
  Background antiretroviral regimen (Efavirenz 600mg QD + Tenofovir 300 mg /Emtricitabine 200 mg QD plus Placebo po BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: maraviroc — Maraviroc 600mg po BID every day from the entry visit until week 48 or until IRIS event or unacceptable toxicity develops.
  Efavirenz 600 mg qd every day from the entry visit until week 48 or until IRIS event or unacceptable toxicity develops.
  Tenofovir/Emtricitabine 300/200 mg qd from the entry visit until week 48 or until IRIS event or unacceptable toxicity develops.
  Other Names: Selzentry; Stocrin; Truvada
  Arms: Maraviroc
Drug: Placebo — Placebo tablets po BID every day from the entry visit until week 48 or until IRIS event or unacceptable toxicity develops.
  Efavirenz 600 mg qd every day from the entry visit until week 48 or until IRIS event or unacceptable toxicity develops.
  Tenofovir/Emtricitabine 300/200 mg qd from the entry visit until week 48 or until IRIS event or unacceptable toxicity develops.
  Other Names: Stocrin; Truvada
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Maraviroc administration can decrease IRIS incidence in HIV infected patients initiating ARV therapy.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo-controlled, multicenter study testing the utility of a CCR5 antagonist (Maraviroc) as an adjuvant to a standard HAART regimen to decrease the incidence of Immune Reconstitution Inflammatory Syndrome (IRIS) in HIV-infected patients naïve to antiretroviral treatment. The study duration will be 60 weeks, 276 subjects (138 per arm) will be recruited. The population included will be HIV-infected patients starting antiretroviral (ARV) therapy at the participating centers in Mexico and South Africa with a CD4 T cell count <100 cells/ul. Subjects will be randomized to receive either Maraviroc (study drug) or placebo in addition to background ARV therapy. The background antiretroviral regimen for all subjects will be: Efavirenz 600mg QD + Tenofovir 300 mg / Emtricitabine 200 mg QD; subjects will be randomized to one of the following arms: Arm A: background ARV + maraviroc 600mg po BID; Arm B: background ARV + placebo po BID. Patients will be followed for 48 weeks. The primary endpoint will be the occurrence of a defined IRIS event by week 24 of follow up. The success of the ARV therapy will also be evaluated by virologic and immunologic response at 24 and 48 weeks. Three immunology sub-studies are planned: 1) Sub-study A will be conformed by a subgroup of 40 subjects (20 from Mexico and 20 from South Africa), additional blood sampling will be performed to evaluate expression of immune activation markers; movement of central memory T cells into cell cycle and frequencies of expandable pathogen-reactive CD4+ and CD8+ T cells in circulation; 2) Sub-study B will be conformed by another subgroup of 60 subjects (all from South Africa), additional blood sampling will be performed to evaluate monocyte and CD4 T cell gene expression as related to activation-induced apoptosis and cytokine secretion.; 3) Sub-study C will evaluate the incidence of thromboembolic disease in the study patients along with baseline evaluation of possible bio-markers of pro-coagulant state.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, as documented by any licensed rapid test kit and confirmed by Western blot or ELISA test kit at any time prior to study enrollment.

Plasma HIV-1 RNA is acceptable as an alternative confirmatory test.

* Men and women age > 18 years.
* Have not received any antiretroviral treatment before entering the study.
* Patients who received Single dose nevirapine or any duration of AZT for PMTC will not be considered ARV naïve.
* CD4+ cell count of </=100 cells/mm3 obtained within 90 days prior to study entry.
* HIV RNA level > 1,000 copies/mL obtained within 90 days prior to study entry.
* Patients with an opportunistic or HIV-related infection may be included according to the clinical judgment of the main investigator in each center when the patient is ready and able to start ARV therapy.
* Laboratory values obtained within 30 days prior to study entry:

  * Absolute neutrophil count (ANC) > 500/mm3.
  * Hemoglobin > 8.0 g/dL.
  * Platelet count > 50,000/mm3.
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase minor of 5 times ULN.
  * Total bilirubin minor of 2.5 times ULN.
  * Creatinine clearance minor of 50* mL/min as estimated by the Cockcroft-Gault equation or Creatinine Clearance > 50ml/min as calculated by a formal creatinine clearance measurement
* All women of reproductive potential (have not reached menopause or undergone hysterectomy, oophorectomy, or tubal ligation) must have a negative serum or urine b-HCG pregnancy test performed within 7 days before study entry.
* Female subjects who are not of reproductive potential (have reached menopause or undergone hysterectomy, oophorectomy, or tubal ligation) or whose male partner has undergone successful vasectomy with resultant azoospermia or has azoospermia for any other reason, are eligible without requiring the use of contraception. Documentation of menopause, sterilization (hysterectomy, oophorectomy, tubal ligation, or vasectomy) and azoospermia by patient-reported history is acceptable.
* All subjects must agree not to participate in a conception process (i.e., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the female study volunteer/male partner must agree to use a form of contraception as specified in the note below while receiving protocol-specified medication(s) and for one month after stopping the medication(s).
* Ability and willingness of subject or legal guardian/representative to give written informed consent.

Exclusion Criteria:

* Pregnancy and breast-feeding.
* Active neoplasia or previous history of neoplasia. (Except localized non visceral Kaposi´s Sarcoma; localized squamous or basal cell carcinoma of the skin, or intraepithelial cervical neoplasia grade III or less).
* Use of the following drugs within 180 days prior to study entry: systemic cancer chemotherapy, systemic investigational agents, and immunomodulators (growth factors, immune globulin, interleukins, interferons).
* Use of systemic corticosteroids in the last 2 weeks prior to randomization.
* Decompensated liver disease (defined as stage C of Child-Pugh classification) at the beginning of the study.
* An altered mental status that in the opinion of the investigator, will compromise the adherence to the protocol.
* Allergy/sensitivity to study drug(s) or their formulations that cannot be substituted by another agent as described in section 5.1
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Serious illness that renders a subject unable to take the antiretroviral study regimen.
* Serious medical illness that in the opinion of the investigator compromises the adherence and/or follow up of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Time to occurrence of an IRIS event | The initial 24 week period of observation

SECONDARY OUTCOMES:
Time to occurrence of a severe IRIS event | The initial 24 week period of observation
Occurrence of either an IRIS event or death | By 24 and 48 weeks
Proportion of subjects who develops an IRIS case | By week 24
Proportion of subjects who develop a severe IRIS case | Week 24
Proportion of subjects who develop a confirmed, non dermatologic IRIS case | Week 24
Proportion of subjects who develop an unmasking or paradoxical IRIS event | Week 24
Frequency of cardiovascular, cerebrovascular, non AIDS related neoplasia, cirrhosis, renal failure and death in both treatment arms | During the study (from entry to week 60)
Frequency of AIDS defining events and AIDS related events in both arms of treatment | From basline to study end
General survival | At week 24 and 48
Survival without IRIS | At weeks 24 and 48
Proportion of patients with VL<50 copies/mL | At weeks 8, 24 and 48
Changes form baseline in CD4+ cells count | From baseline to weeks 12, 24 and 48
Safety and tolerability of the treatment regimens | Along the study
Incidence of HIV drug resistance | Baseline to week 60
Prevalence of CCR5 tropism | Baseline
Prevalence of CCR5 HIV tropism | At virological failure occurrence
Baseline predictors of IRIS | Baseline
Genetic polymorphisms associated with the occurrence of IRIS | Baseline
To evaluate the rol of biomarkers (CRP) in predicting or identifying IRIS and the effect of Maraviroc on this marker | Baseline to IRIS event

CONTACTS AND LOCATIONS:
Overall Officials: Ian Sanne, MBBCH, FCP, Principal Investigator — University of the Witwatersrand. Themba Lethu Clinic.; Michael M. Lederman, MD, Principal Investigator — Center for AIDS Research. Case Western Reserve University; Luis J Montaner, M.Sc., Principal Investigator — HIV-1 Immunopathogenesis Laboratory. The Wistar Institute; Livio Azzoni, MD, PhD, Principal Investigator — HIV-1 Immunopathogenesis Laboratory. The Wistar Institute; Juan G Sierra Madero, MD, Principal Investigator — Insituto Nacional de Nutricion de Ciencias Medicas y Nutricion Salvador Zubiran; Susan Ellenberg, Ph.D., Principal Investigator — Center for Clinical Epidemiology and Biostatistics, University of Pennsylvania School of Medicine; Irini Sereti, M.D., MHS, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (10):
- United States (4):
  - NIH/NIAD, Bethesda, Maryland
  - Center for AIDS Research. Case Western Reserve University, Cleveland, Ohio
  - Center for Clinical Epidemiology and Biostatistics. University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - HIV-1 Immunopathogenesis Laboratory. The Wistar Institute, Philadelphia, Pennsylvania
- Mexico (5):
  - Hospital General de León, León, Guanajuato
  - Hospital Civil de Guadalajara, Guadalajara, Jalisco
  - Hospital General de México, Mexico City, Mexico City
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City
  - Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí
- Clinical HIV Research Unit. Themba Lethu Clinic. Helen Joseph Hospital, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Background] Jensen-Fangel S, Pedersen L, Pedersen C, Larsen CS, Tauris P, Moller A, Sorensen HT, Obel N. Low mortality in HIV-infected patients starting highly active antiretroviral therapy: a comparison with the general population. AIDS. 2004 Jan 2;18(1):89-97. doi: 10.1097/00002030-200401020-00011. PMID 15090834
- [Background] Corey DM, Kim HW, Salazar R, Illescas R, Villena J, Gutierrez L, Sanchez J, Tabet SR. Brief report: effectiveness of combination antiretroviral therapy on survival and opportunistic infections in a developing world setting: an observational cohort study. J Acquir Immune Defic Syndr. 2007 Apr 1;44(4):451-5. doi: 10.1097/QAI.0b013e31802f8512. PMID 17195766
- [Background] Lederman MM. Immune restoration and CD4+ T-cell function with antiretroviral therapies. AIDS. 2001 Feb;15 Suppl 2:S11-5. doi: 10.1097/00002030-200102002-00003. PMID 11424971
- [Background] Lawn SD, Myer L, Bekker LG, Wood R. CD4 cell count recovery among HIV-infected patients with very advanced immunodeficiency commencing antiretroviral treatment in sub-Saharan Africa. BMC Infect Dis. 2006 Mar 21;6:59. doi: 10.1186/1471-2334-6-59. PMID 16551345
- [Background] Battegay M, Nuesch R, Hirschel B, Kaufmann GR. Immunological recovery and antiretroviral therapy in HIV-1 infection. Lancet Infect Dis. 2006 May;6(5):280-7. doi: 10.1016/S1473-3099(06)70463-7. PMID 16631548
- [Background] Murdoch DM, Venter WD, Van Rie A, Feldman C. Immune reconstitution inflammatory syndrome (IRIS): review of common infectious manifestations and treatment options. AIDS Res Ther. 2007 May 8;4:9. doi: 10.1186/1742-6405-4-9. PMID 17488505
- [Background] Autran B, Carcelain G, Li TS, Blanc C, Mathez D, Tubiana R, Katlama C, Debre P, Leibowitch J. Positive effects of combined antiretroviral therapy on CD4+ T cell homeostasis and function in advanced HIV disease. Science. 1997 Jul 4;277(5322):112-6. doi: 10.1126/science.277.5322.112. PMID 9204894
- [Background] Shelburne SA, Visnegarwala F, Darcourt J, Graviss EA, Giordano TP, White AC Jr, Hamill RJ. Incidence and risk factors for immune reconstitution inflammatory syndrome during highly active antiretroviral therapy. AIDS. 2005 Mar 4;19(4):399-406. doi: 10.1097/01.aids.0000161769.06158.8a. PMID 15750393
- [Background] Lederman MM, Penn-Nicholson A, Cho M, Mosier D. Biology of CCR5 and its role in HIV infection and treatment. JAMA. 2006 Aug 16;296(7):815-26. doi: 10.1001/jama.296.7.815. PMID 16905787
- [Background] Westby M, van der Ryst E. CCR5 antagonists: host-targeted antivirals for the treatment of HIV infection. Antivir Chem Chemother. 2005;16(6):339-54. doi: 10.1177/095632020501600601. PMID 16329283
- [Background] Knobel H, Alonso J, Casado JL, Collazos J, Gonzalez J, Ruiz I, Kindelan JM, Carmona A, Juega J, Ocampo A; GEEMA Study Group. Validation of a simplified medication adherence questionnaire in a large cohort of HIV-infected patients: the GEEMA Study. AIDS. 2002 Mar 8;16(4):605-13. doi: 10.1097/00002030-200203080-00012. PMID 11873004
- [Background] French MA, Lenzo N, John M, Mallal SA, McKinnon EJ, James IR, Price P, Flexman JP, Tay-Kearney ML. Immune restoration disease after the treatment of immunodeficient HIV-infected patients with highly active antiretroviral therapy. HIV Med. 2000 Mar;1(2):107-15. doi: 10.1046/j.1468-1293.2000.00012.x. PMID 11737333
- [Background] Jevtovic DJ, Salemovic D, Ranin J, Pesic I, Zerjav S, Djurkovic-Djakovic O. The prevalence and risk of immune restoration disease in HIV-infected patients treated with highly active antiretroviral therapy. HIV Med. 2005 Mar;6(2):140-3. doi: 10.1111/j.1468-1293.2005.00277.x. PMID 15807721
- [Background] French MA, Price P, Stone SF. Immune restoration disease after antiretroviral therapy. AIDS. 2004 Aug 20;18(12):1615-27. doi: 10.1097/01.aids.0000131375.21070.06. PMID 15280772
- [Background] Singh N, Perfect JR. Immune reconstitution syndrome associated with opportunistic mycoses. Lancet Infect Dis. 2007 Jun;7(6):395-401. doi: 10.1016/S1473-3099(07)70085-3. PMID 17521592
- [Background] Bonnet MM, Pinoges LL, Varaine FF, Oberhauser BB, O'Brien DD, Kebede YY, Hewison CC, Zachariah RR, Ferradini LL. Tuberculosis after HAART initiation in HIV-positive patients from five countries with a high tuberculosis burden. AIDS. 2006 Jun 12;20(9):1275-9. doi: 10.1097/01.aids.0000232235.26630.ee. PMID 16816556
- [Background] Rodriguez-Rosado R, Soriano V, Dona C, Gonzalez-Lahoz J. Opportunistic infections shortly after beginning highly active antiretroviral therapy. Antivir Ther. 1998;3(4):229-31. PMID 10682143
- [Background] Lortholary O, Fontanet A, Memain N, Martin A, Sitbon K, Dromer F; French Cryptococcosis Study Group. Incidence and risk factors of immune reconstitution inflammatory syndrome complicating HIV-associated cryptococcosis in France. AIDS. 2005 Jul 1;19(10):1043-9. doi: 10.1097/01.aids.0000174450.70874.30. PMID 15958835
- [Background] Michelet C, Arvieux C, Francois C, Besnier JM, Rogez JP, Breux JP, Souala F, Allavena C, Raffi F, Garre M, Cartier F. Opportunistic infections occurring during highly active antiretroviral treatment. AIDS. 1998 Oct 1;12(14):1815-22. doi: 10.1097/00002030-199814000-00013. PMID 9792382
- [Background] Park WB, Choe PG, Jo JH, Kim SH, Bang JH, Kim HB, Kim NJ, Oh MD, Choe KW. Tuberculosis manifested by immune reconstitution inflammatory syndrome during HAART. AIDS. 2007 Apr 23;21(7):875-7. doi: 10.1097/QAD.0b013e3280f7751f. PMID 17415046
- [Background] Domingo P, Torres OH, Ris J, Vazquez G. Herpes zoster as an immune reconstitution disease after initiation of combination antiretroviral therapy in patients with human immunodeficiency virus type-1 infection. Am J Med. 2001 Jun 1;110(8):605-9. doi: 10.1016/s0002-9343(01)00703-3. PMID 11382367
- [Background] Manosuthi W, Kiertiburanakul S, Phoorisri T, Sungkanuparph S. Immune reconstitution inflammatory syndrome of tuberculosis among HIV-infected patients receiving antituberculous and antiretroviral therapy. J Infect. 2006 Dec;53(6):357-63. doi: 10.1016/j.jinf.2006.01.002. Epub 2006 Feb 17. PMID 16487593
- [Background] Madec Y, Laureillard D, Pinoges L, Fernandez M, Prak N, Ngeth C, Moeung S, Song S, Balkan S, Ferradini L, Quillet C, Fontanet A. Response to highly active antiretroviral therapy among severely immuno-compromised HIV-infected patients in Cambodia. AIDS. 2007 Jan 30;21(3):351-9. doi: 10.1097/QAD.0b013e328012c54f. PMID 17255742
- [Background] Braitstein P, Brinkhof MW, Dabis F, Schechter M, Boulle A, Miotti P, Wood R, Laurent C, Sprinz E, Seyler C, Bangsberg DR, Balestre E, Sterne JA, May M, Egger M; Antiretroviral Therapy in Lower Income Countries (ART-LINC) Collaboration; ART Cohort Collaboration (ART-CC) groups. Mortality of HIV-1-infected patients in the first year of antiretroviral therapy: comparison between low-income and high-income countries. Lancet. 2006 Mar 11;367(9513):817-24. doi: 10.1016/S0140-6736(06)68337-2. PMID 16530575
- [Background] Zachariah R, Fitzgerald M, Massaquoi M, Pasulani O, Arnould L, Makombe S, Harries AD. Risk factors for high early mortality in patients on antiretroviral treatment in a rural district of Malawi. AIDS. 2006 Nov 28;20(18):2355-60. doi: 10.1097/QAD.0b013e32801086b0. PMID 17117022
- [Background] Sabin CA, Smith CJ, Gumley H, Murphy G, Lampe FC, Phillips AN, Prinz B, Youle M, Johnson MA. Late presenters in the era of highly active antiretroviral therapy: uptake of and responses to antiretroviral therapy. AIDS. 2004 Nov 5;18(16):2145-51. doi: 10.1097/00002030-200411050-00006. PMID 15577647
- [Background] Manabe YC, Campbell JD, Sydnor E, Moore RD. Immune reconstitution inflammatory syndrome: risk factors and treatment implications. J Acquir Immune Defic Syndr. 2007 Dec 1;46(4):456-62. doi: 10.1097/qai.0b013e3181594c8c. PMID 18077835
- [Background] Lawn SD, Myer L, Bekker LG, Wood R. Tuberculosis-associated immune reconstitution disease: incidence, risk factors and impact in an antiretroviral treatment service in South Africa. AIDS. 2007 Jan 30;21(3):335-41. doi: 10.1097/QAD.0b013e328011efac. PMID 17255740
- [Background] Delves PJ, Roitt IM. The immune system. First of two parts. N Engl J Med. 2000 Jul 6;343(1):37-49. doi: 10.1056/NEJM200007063430107. No abstract available. PMID 10882768
- [Background] Palella FJ Jr, Delaney KM, Moorman AC, Loveless MO, Fuhrer J, Satten GA, Aschman DJ, Holmberg SD. Declining morbidity and mortality among patients with advanced human immunodeficiency virus infection. HIV Outpatient Study Investigators. N Engl J Med. 1998 Mar 26;338(13):853-60. doi: 10.1056/NEJM199803263381301. PMID 9516219
- [Background] Egger M, Hirschel B, Francioli P, Sudre P, Wirz M, Flepp M, Rickenbach M, Malinverni R, Vernazza P, Battegay M. Impact of new antiretroviral combination therapies in HIV infected patients in Switzerland: prospective multicentre study. Swiss HIV Cohort Study. BMJ. 1997 Nov 8;315(7117):1194-9. doi: 10.1136/bmj.315.7117.1194. PMID 9393221
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] Storey JD, Tibshirani R. Statistical significance for genomewide studies. Proc Natl Acad Sci U S A. 2003 Aug 5;100(16):9440-5. doi: 10.1073/pnas.1530509100. Epub 2003 Jul 25. PMID 12883005
- [Background] Lederman MM, Margolis L. The lymph node in HIV pathogenesis. Semin Immunol. 2008 Jun;20(3):187-95. doi: 10.1016/j.smim.2008.06.001. Epub 2008 Jul 14. PMID 18620868
- [Background] Sieg SF, Bazdar DA, Lederman MM. S-phase entry leads to cell death in circulating T cells from HIV-infected persons. J Leukoc Biol. 2008 Jun;83(6):1382-7. doi: 10.1189/jlb.0907643. Epub 2008 Mar 27. PMID 18372341
- [Background] Sieg SF, Rodriguez B, Asaad R, Jiang W, Bazdar DA, Lederman MM. Peripheral S-phase T cells in HIV disease have a central memory phenotype and rarely have evidence of recent T cell receptor engagement. J Infect Dis. 2005 Jul 1;192(1):62-70. doi: 10.1086/430620. Epub 2005 May 26. PMID 15942895
- [Background] Brenchley JM, Price DA, Schacker TW, Asher TE, Silvestri G, Rao S, Kazzaz Z, Bornstein E, Lambotte O, Altmann D, Blazar BR, Rodriguez B, Teixeira-Johnson L, Landay A, Martin JN, Hecht FM, Picker LJ, Lederman MM, Deeks SG, Douek DC. Microbial translocation is a cause of systemic immune activation in chronic HIV infection. Nat Med. 2006 Dec;12(12):1365-71. doi: 10.1038/nm1511. Epub 2006 Nov 19. PMID 17115046
- [Background] Jiang W, Lederman MM, Hunt P, Sieg SF, Haley K, Rodriguez B, Landay A, Martin J, Sinclair E, Asher AI, Deeks SG, Douek DC, Brenchley JM. Plasma levels of bacterial DNA correlate with immune activation and the magnitude of immune restoration in persons with antiretroviral-treated HIV infection. J Infect Dis. 2009 Apr 15;199(8):1177-85. doi: 10.1086/597476. PMID 19265479
- [Background] Funderburg N, Luciano AA, Jiang W, Rodriguez B, Sieg SF, Lederman MM. Toll-like receptor ligands induce human T cell activation and death, a model for HIV pathogenesis. PLoS One. 2008 Apr 2;3(4):e1915. doi: 10.1371/journal.pone.0001915. PMID 18382686
- [Background] Pandrea I, Apetrei C, Gordon S, Barbercheck J, Dufour J, Bohm R, Sumpter B, Roques P, Marx PA, Hirsch VM, Kaur A, Lackner AA, Veazey RS, Silvestri G. Paucity of CD4+CCR5+ T cells is a typical feature of natural SIV hosts. Blood. 2007 Feb 1;109(3):1069-76. doi: 10.1182/blood-2006-05-024364. Epub 2006 Sep 26. PMID 17003371
- [Background] Bourgarit A, Carcelain G, Martinez V, Lascoux C, Delcey V, Gicquel B, Vicaut E, Lagrange PH, Sereni D, Autran B. Explosion of tuberculin-specific Th1-responses induces immune restoration syndrome in tuberculosis and HIV co-infected patients. AIDS. 2006 Jan 9;20(2):F1-7. doi: 10.1097/01.aids.0000202648.18526.bf. PMID 16511406
- [Background] Salkowitz JR, Sieg SF, Harding CV, Lederman MM. In vitro human memory CD8 T cell expansion in response to cytomegalovirus requires CD4+ T cell help. J Infect Dis. 2004 Mar 15;189(6):971-83. doi: 10.1086/382032. Epub 2004 Mar 1. PMID 14999599
- [Background] Ratnam I, Chiu C, Kandala NB, Easterbrook PJ. Incidence and risk factors for immune reconstitution inflammatory syndrome in an ethnically diverse HIV type 1-infected cohort. Clin Infect Dis. 2006 Feb 1;42(3):418-27. doi: 10.1086/499356. Epub 2005 Dec 28. PMID 16392092
- [Derived] Araujo-Pereira M, Barreto-Duarte B, Arriaga MB, Musselwhite LW, Vinhaes CL, Belaunzaran-Zamudio PF, Rupert A, Montaner LJ, Lederman MM, Sereti I, Madero JGS, Andrade BB. Relationship Between Anemia and Systemic Inflammation in People Living With HIV and Tuberculosis: A Sub-Analysis of the CADIRIS Clinical Trial. Front Immunol. 2022 Jun 23;13:916216. doi: 10.3389/fimmu.2022.916216. eCollection 2022. PMID 35812431
- [Derived] Sierra-Madero JG, Ellenberg SS, Rassool MS, Tierney A, Belaunzaran-Zamudio PF, Lopez-Martinez A, Pineirua-Menendez A, Montaner LJ, Azzoni L, Benitez CR, Sereti I, Andrade-Villanueva J, Mosqueda-Gomez JL, Rodriguez B, Sanne I, Lederman MM; CADIRIS study team. Effect of the CCR5 antagonist maraviroc on the occurrence of immune reconstitution inflammatory syndrome in HIV (CADIRIS): a double-blind, randomised, placebo-controlled trial. Lancet HIV. 2014 Nov;1(2):e60-7. doi: 10.1016/S2352-3018(14)70027-X. Epub 2014 Oct 21. PMID 26423989
- [Derived] Sierra-Madero JG, Ellenberg S, Rassool MS, Tierney A, Belaunzaran-Zamudio PF, Lopez-Martinez A, Pineirua-Menendez A, Montaner LJ, Azzoni L, Benitez CR, Sereti I, Andrade-Villanueva J, Mosqueda-Gomez JL, Rodriguez B, Sanne I, Lederman MM; CADIRIS study team. A Randomized, Double-Blind, Placebo-Controlled Clinical Trial of a Chemokine Receptor 5 (CCR5) Antagonist to Decrease the Occurrence of Immune Reconstitution Inflammatory Syndrome in HIV-Infection: The CADIRIS Study. Lancet HIV. 2014 Nov 1;1(2):e60-e67. doi: 10.1016/S2352-3018(14)70027-X. PMID 26366430